CLINICAL TRIAL: NCT01193244
Title: A Phase 3, Randomized, Double-Blind, Multicenter Trial Comparing Orteronel Plus Prednisone With Placebo Plus Prednisone in Patients With Chemotherapy-Naive Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study Comparing Orteronel Plus Prednisone in Participants With Chemotherapy-Naive Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C21004; 2010-018661-35 (EudraCT Number); 0991413276 (Other: TCTIP); 10/H0406/75 (Registry Identifier: NRES); U1111-1181-0387 (Registry Identifier: WHO)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Orteronel + prednisone (Experimental)
  Interventions: Drug: Orteronel; Drug: Prednisone
- Placebo + prednisone (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Prednisone

INTERVENTIONS:
Drug: Orteronel — Orteronel will be administered orally twice a day continuously throughout the study. Patients will also receive concomitant gonadotropin-releasing hormone (GnRH) analogue therapy unless they have previously undergone orchiectomy and have a testosterone concentration of <50 ng/dL.
  Arms: Orteronel + prednisone
Drug: Placebo — Placebo will be administered orally twice a day continuously throughout the study. Additionally, all patients will receive concomitant gonadotropin-releasing hormone (GnRH) analogue therapy unless they have previously undergone orchiectomy and a testosterone concentration of <50 ng/dL.
  Arms: Placebo + prednisone
Drug: Prednisone — Prednisone will be administered orally twice a day continuously throughout the study. Patients will also receive concomitant gonadotropin-releasing hormone (GnRH) analogue therapy unless they have previously undergone orchiectomy and have a testosterone concentration of <50 ng/dL.

SUMMARY:
This is a randomized, double-blind, multicenter, phase 3 study evaluating orteronel (TAK-700) plus prednisone compared with placebo plus prednisone in the treatment of men with progressive, chemotherapy-naive, metastatic, castration-resistant prostate cancer (mCRPC)

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria:

* Voluntary written consent
* Male patients 18 years or older
* Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma
* Radiograph-documented metastatic disease
* Progressive disease
* Prior surgical castration or concurrent use of an agent for medical castration
* Either absence of pain or pain not requiring use of any opioid or narcotic analgesia in the 2 weeks prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Even if surgically sterilized, patients must practice effective barrier contraception during the entire study treatment and for 4 months after the last dose of study drug, OR abstain from heterosexual intercourse
* Meet screening laboratory values as specified in protocol
* Stable medical condition

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Known hypersensitivity to orteronel, prednisone or gonadotropin-releasing hormone (GnRH) analogue
* Received prior therapy with orteronel, aminoglutethimide, ketoconazole or abiraterone
* Received antiandrogen therapy within 6 weeks for bicalutamide and 4 weeks for all others prior to first dose of study drug
* Continuous daily use of oral prednisone or oral dexamethasone for more than 14 days within 3 months prior to study
* Received prior chemotherapy for prostate cancer with exception of neoadjuvant/adjuvant therapy as part of initial primary treatment for local disease that was completed 2 or more years prior to screening
* Exposure to radioisotope therapy within 4 weeks of receiving first dose of study drug; exposure to external beam radiation within 2 weeks of start of screening until receiving the first dose of study drug
* Documented central nervous system metastases
* Treatment with any investigational compound within 30 days prior to first dose of study drug
* Current spinal cord compression, bilateral hydronephrosis or current bladder neck outlet obstruction
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Uncontrolled cardiovascular condition as specified in study protocol
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Unwilling or unable to comply with protocol
* Uncontrolled nausea, vomiting or diarrhea
* Known gastrointestinal disease or procedure that could interfere with oral absorption or tolerance of orteronel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (240):
- United States (48):
  - Anchorage, Alaska
  - Tucson, Arizona
  - Duarte, California
  - Highland, California
  - Orange, California
  - Sacramento, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - Deerfield Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Port Saint Lucie, Florida
  - Jeffersonville, Indiana
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Lansing, Michigan
  - Duluth, Minnesota
  - Corinth, Mississippi
  - Columbia, Missouri
  - Jefferson City, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - East Syracuse, New York
  - New York, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Kettering, Ohio
  - Tualatin, Oregon
  - Hershey, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Piitsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Denton, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Australia (7):
  - Garran
  - Hobart
  - Kurralta Park
  - Nedlands
  - Perth
  - Redcliffe
  - Wodonga
- Austria (3):
  - Graz
  - Linz
  - Vienna
- Minsk, Belarus
- Belgium (5):
  - Edegem
  - Hasselt
  - Kortrijk
  - Leuven
  - Namur
- Brazil (21):
  - Bairro Nazare - Salvador
  - Barretos/sp
  - Belo Horizonte
  - Campinas
  - Caxias do Sul
  - Curitiba
  - Fortaleza/ce
  - Ijuí
  - Joinville
  - Lajeado - Rs
  - Piracicaba - Sp
  - Porto Alegre- Rs
  - Porto Alegre/rs
  - Ribeirao Preto - Sp
  - Rio de Janeiro
  - Rio de Janeiro Rj
  - Santo André
  - São José do Rio Preto
  - São José dos Campos
  - São Paulo
  - Sorocaba - Sp
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Canada (10):
  - Kelowna, British Columbia
  - Burlington, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Owen Sound, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- Chile (4):
  - Las Condes
  - Santiago
  - Temuco
  - Valparaíso
- Cali, Colombia
- Czechia (2):
  - Hradec Králové
  - Prague
- Finland (4):
  - Joensuu
  - Oulu
  - Seinäjoki
  - Tampere
- France (13):
  - Angers
  - Bordeaux
  - Caen
  - Créteil
  - La Roche-sur-Yon
  - Lyon
  - Marseille
  - Nancy
  - Nantes
  - Paris
  - Poitiers
  - Saint-Etienne
  - Villejuif
- Germany (9):
  - Braunschweig
  - Dresden
  - Hamburg
  - Hanover
  - Kassel
  - Kempen
  - Nürtingen
  - Tübingen
  - Wuppertal
- Greece (5):
  - Athens
  - Heraklion Crete
  - Larissa
  - Pátrai
  - Thessaloniki
- Hong Kong (2):
  - Kowloon
  - Shatin
- Ireland (2):
  - Dublin
  - Galway
- Israel (7):
  - Haifa
  - Holon
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Italy (4):
  - Aviano
  - Novara
  - Roma
  - Torino
- Japan (18):
  - Chiba
  - Fukuoka
  - Hamamatsu
  - Hokkaido
  - Kanazawa
  - Kita-gun
  - Maebashi
  - Mito
  - Osaka
  - Sakura
  - Sayama
  - Sendai
  - Shimizucho Sunto-gun
  - Suntou-gun
  - Tokyo
  - Yamagata
  - Yokohama
  - Yufu
- Riga, Latvia
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Mexico (3):
  - Durango Durango
  - Mexico City Distrito Federal
  - Zapopan Jalisco
- Netherlands (8):
  - Amsterdam
  - Arnhem
  - Breda
  - Eindhoven
  - Heerlen
  - Nieuwegein
  - Nijmegen
  - Rotterdam
- New Zealand (5):
  - Auckland
  - Christchurch
  - Dunedin
  - Takapuna
  - Tauranga
- Lima, Peru
- Poland (2):
  - Bielsko-Biala
  - Wroclaw
- Portugal (3):
  - Liepaja
  - Lisbon
  - Porto
- San Juan, PR, Puerto Rico
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (2):
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Slovakia (4):
  - Nitra
  - Prešov
  - Trenčín
  - Žilina
- South Africa (4):
  - Cape Town
  - Durban
  - George
  - Port Elizabeth
- Spain (7):
  - A Coruña
  - Barcelona
  - Madrid
  - Majadahonda
  - Pamplona
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala
- Switzerland (4):
  - Aarau
  - Lausanne
  - Winterthur
  - Zurich
- Taiwan (2):
  - Taichung
  - Taipei
- Ukraine (4):
  - Dnipropetrovsk
  - Donetsk
  - Kyiv
  - Zaporizhzhya
- United Kingdom (11):
  - Aberdeen
  - Belfast
  - Bristol
  - Cottingham
  - Coventry
  - Glasgow
  - London
  - Manchester
  - Northwood
  - Preston
  - Southampton

REFERENCES:
- [Derived] Heller G, McCormack R, Kheoh T, Molina A, Smith MR, Dreicer R, Saad F, de Wit R, Aftab DT, Hirmand M, Limon A, Fizazi K, Fleisher M, de Bono JS, Scher HI. Circulating Tumor Cell Number as a Response Measure of Prolonged Survival for Metastatic Castration-Resistant Prostate Cancer: A Comparison With Prostate-Specific Antigen Across Five Randomized Phase III Clinical Trials. J Clin Oncol. 2018 Feb 20;36(6):572-580. doi: 10.1200/JCO.2017.75.2998. Epub 2017 Dec 22. PMID 29272162
- [Derived] Suri A, Chapel S, Lu C, Venkatakrishnan K. Physiologically based and population PK modeling in optimizing drug development: A predict-learn-confirm analysis. Clin Pharmacol Ther. 2015 Sep;98(3):336-44. doi: 10.1002/cpt.155. Epub 2015 Jul 14. PMID 26031410
- [Derived] Saad F, Fizazi K, Jinga V, Efstathiou E, Fong PC, Hart LL, Jones R, McDermott R, Wirth M, Suzuki K, MacLean DB, Wang L, Akaza H, Nelson J, Scher HI, Dreicer R, Webb IJ, de Wit R; ELM-PC 4 investigators. Orteronel plus prednisone in patients with chemotherapy-naive metastatic castration-resistant prostate cancer (ELM-PC 4): a double-blind, multicentre, phase 3, randomised, placebo-controlled trial. Lancet Oncol. 2015 Mar;16(3):338-48. doi: 10.1016/S1470-2045(15)70027-6. Epub 2015 Feb 18. PMID 25701170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 324 investigative sites in North America, Europe, Australia, Brazil, Chile, Colombia, Hong Kong, Peru, Puerto Rico, Israel, Japan, Mexico, New Zealand, Singapore, South Africa, and Taiwan from 19 October 2010 to 7 April 2016.
Pre-assignment Details: Male participants who were chemotherapy-naive and had metastatic castration-resistant prostate cancer (mCRPC) with documented progressive metastatic disease were enrolled in 1 of 2 treatment groups to receive Orteronel 400 milligram (mg) + Prednisone 5 mg or Placebo + Prednisone 5 mg.
Groups:
- Placebo + Prednisone 5 mg: Orteronel placebo-matching tablets, orally, twice daily (BID) and Prednisone 5 mg, tablets, orally, BID for up to Day 28 of each treatment cycle throughout the study.
- Orteronel 400 mg + Prednisone 5 mg: Orteronel 400 mg, tablets, orally, BID and Prednisone 5 mg, tablets, orally, BID for up to Day 28 of each treatment cycle throughout the study. In Japan, participants were administered with Orteronel 300 mg, tablets, orally, BID and Prednisone 5 mg, tablets, orally, BID for up to Day 28 of each treatment cycle throughout the study.
Period: Overall Study
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Started | 779 | 781
Treated | 770 (Participants who continued to receive Placebo after unblinding.) | 784 (Participants randomized to receive Placebo but crossed-over to receive Orteronel after unblinding.)
Completed | 391 | 391
Not Completed | 388 | 390
Not completed — Withdrawal by Subject | 79 | 97
Not completed — Other | 303 | 278
Not completed — Lost to Follow-up | 6 | 15

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg | Total
Number analyzed (Participants) | 779 | 781 | 1560
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.19) | 70.9 (8.26) | 71.0 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 779 | 781 | 1560
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 90 | 107 | 197
  Not Hispanic or Latino | 672 | 669 | 1341
  Unknown or Not Reported | 17 | 5 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 10 | 12 | 22
  Asian | 51 | 38 | 89
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 19 | 25 | 44
  White | 670 | 685 | 1355
  Unknown or Not Reported | 12 | 3 | 15
  Other | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 22 | 44
  United States | 147 | 148 | 295
  Austria | 12 | 12 | 24
  Belarus | 6 | 10 | 16
  Belgium | 18 | 21 | 39
  Bulgaria | 6 | 6 | 12
  Croatia | 5 | 1 | 6
  Czech Republic | 13 | 18 | 31
  Estonia | 2 | 4 | 6
  Finland | 9 | 4 | 13
  France | 66 | 55 | 121
  Germany | 29 | 40 | 69
  Greece | 23 | 16 | 39
  Hungary | 3 | 4 | 7
  Ireland | 11 | 13 | 24
  Italy | 10 | 8 | 18
  Latvia | 12 | 14 | 26
  Lithuania | 19 | 18 | 37
  Netherlands | 35 | 38 | 73
  Poland | 0 | 4 | 4
  Portugal | 4 | 4 | 8
  Romania | 20 | 13 | 33
  Slovakia | 9 | 11 | 20
  Spain | 14 | 12 | 26
  Sweden | 11 | 6 | 17
  Switzerland | 10 | 8 | 18
  Ukraine | 25 | 23 | 48
  United Kingdom | 42 | 53 | 95
  Australia | 27 | 27 | 54
  Brazil | 41 | 50 | 91
  Chile | 20 | 20 | 40
  Colombia | 3 | 6 | 9
  Hong Kong | 1 | 3 | 4
  Israel | 14 | 4 | 18
  Japan | 22 | 18 | 40
  Mexico | 7 | 9 | 16
  New Zealand | 25 | 26 | 51
  Peru | 6 | 10 | 16
  Puerto Rico | 1 | 1 | 2
  Singapore | 5 | 2 | 7
  South Africa | 6 | 4 | 10
  Taiwan, Province Of China | 12 | 10 | 22
  Russia | 6 | 5 | 11
Height [Mean (Standard Deviation); unit: centimeter] — Height data was available for 1558 participants as follows: n= 778, 780.
  centimeter | 172.77 (7.485) | 173.26 (7.858) | 173.02 (7.675)
Weight [Mean (Standard Deviation); unit: kilogram] — Weight data was available for 1559 participants as follows: n= 778, 781.
  kilogram | 84.04 (15.846) | 85.09 (16.286) | 84.57 (16.071)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI data was available for 1557 participants as follows: n= 777, 780.
  kilogram per square meter (kg/m^2) | 28.09 (4.651) | 28.28 (4.730) | 28.19 (4.690)

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: rPFS was defined as the time from randomization to the first objective evidence of radiographic disease progression assessed by independent central radiology review or death due to any cause, whichever occurred first. Radiographic disease progression was evaluated by computerized tomography (CT) scan or magnetic resonance imaging (MRI) and radionuclide bone scans at regularly scheduled visits. Radiographic disease progression in bone required a confirmatory scan. Radiographic disease progression in soft tissue did not require a confirmatory scan for purposes of analysis. Radiographic disease progression was evaluated by independent central radiology review using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 for soft tissue disease and Prostate Cancer Working Group (PCWG2) guidelines for bone disease. Participants who did not reach the endpoint were censored at their last assessment.
Time Frame: Baseline until radiographic disease progression or death, whichever occurred first (approximately up to 4.7 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 8.7 [8.32 to 10.91] | 13.8 [13.05 to 14.92]
Statistical Analysis 1: Comparison: Placebo + Prednisone 5 mg vs Orteronel 400 mg + Prednisone 5 mg; Hazard ratio is based on a stratified Cox's proportional hazard regression model with stratification factors of region and radiographic disease progression at baseline with treatment as a factor in the model. A hazard ratio less than (<) 1 indicated better prevention of death in the orteronel group compared to the placebo group. From log-rank test stratified by region and radiographic disease progression at Baseline; Test type: Superiority or Other; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.707, 95% CI [0.626 to 0.799]

2. Primary Outcome: Overall Survival
Description: Overall survival was calculated from the date of participant randomization to the date of participant death due to any cause. Participants without documentation of death at time of the analysis were censored as of the date the participant was last known to be alive, or the data cutoff date, whichever was earlier.
Time Frame: Baseline until death (up to 4.7 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 29.5 [27.28 to 32.38] | 29.9 [27.88 to 33.04]
Statistical Analysis 1: Comparison: Placebo + Prednisone 5 mg vs Orteronel 400 mg + Prednisone 5 mg; Hazard ratio is based on a stratified Cox's proportional hazard regression model with stratification factors of region and radiographic disease progression at baseline with treatment as a factor in the model. A hazard ratio <1 indicated better prevention of death in the orteronel group compared to the placebo group. From log-rank test stratified by region and radiographic disease progression at baseline; Test type: Superiority or Other; p = 0.59755, Log Rank; Hazard Ratio (HR) = 0.963, 95% CI [0.838 to 1.107]

3. Secondary Outcome: Percentage of Participants Achieving 50 Percent Reduction From Baseline in Prostate Specific Antigen (PSA50) Response at Week 12
Description: The PSA50 is defined as a decline of at least 50 percent (%) from baseline.
Time Frame: Week 12
Population: ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
percentage of participants | 24.6 [21.7 to 27.8] | 42.6 [39.1 to 46.2]
Statistical Analysis 1: Comparison: Placebo + Prednisone 5 mg vs Orteronel 400 mg + Prednisone 5 mg; Logistic regression model with prognostic factors: region; radiographic disease progression at baseline; age; race; baseline Eastern Cooperative Oncology Group (ECOG) score; Gleason score at initial diagnosis; baseline PSA, natural log scale; presence of visceral disease; alkaline phosphatase; lactate dehydrogenase; and hemoglobin. Odds ratio greater than (>)1 favored orteronel. P-values tested for odds ratio equal to 1; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.166, 95% CI [1.724 to 2.721]

4. Secondary Outcome: Percentage of Participants With Favorable Circulating Tumor Cell Count (CTC) Levels at Week 12
Description: A favorable CTC count was defined as less than <5 counts per 7.5 milliliter (mL) in whole blood. An unfavorable CTC count was defined as greater than or equal to (>=) 5 counts/7.5 mL in whole blood.
Time Frame: Week 12
Population: ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
percentage of participants | 9.1 [7.2 to 11.4] | 15.4 [12.9 to 18.1]
Statistical Analysis 1: Comparison: Placebo + Prednisone 5 mg vs Orteronel 400 mg + Prednisone 5 mg; Logistic regression model with prognostic factors: region; radiographic disease progression at baseline; age; race; baseline ECOG score; Gleason score at initial diagnosis; baseline PSA, natural log scale; presence of visceral disease; alkaline phosphatase; lactate dehydrogenase; and hemoglobin. Odds ratio > 1 favored orteronel. P-values tested for odds ratio equal to 1; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.712, 95% CI [1.235 to 2.373]

5. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time from participant randomization to the first assessment date of pain progression. Pain progression was defined as the occurrence of 1 of the following and confirmed by an additional assessment, at least 3 weeks but not more than 5 weeks later: The brief pain inventory-short form (BPI-SF) worst pain score was >=4 with a >=2 point increase over baseline in BPI-SF worst pain score with stable or increased analgesic use; The BPI-SF worst pain score was >=4 but not less than baseline with new or increased (relative to baseline) Step II or Step III analgesic use; The BPI-SF worst pain score was <=3 but not less than baseline with new or increased (relative to baseline) Step III analgesic use. BPI-SF was an 11-item questionnaire, designed to assess severity and impact of pain on daily functions. Total score ranged from 0 to 100 with lower scores being indicative of less pain or pain interference.
Time Frame: Baseline until End of treatment (EOT) (approximately up to 4.7 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | NA [NA to NA] — Median was not estimable due to low number of events in the arm. | NA [28.57 to NA] — Median was not estimable due to low number of events in the arm.
Statistical Analysis 1: Comparison: Placebo + Prednisone 5 mg vs Orteronel 400 mg + Prednisone 5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.33906, Log Rank; Hazard Ratio (HR) = 0.885, 95% CI [0.688 to 1.138]

6. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 61 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 770 | 784
participants
  TEAE | 733 | 769
  Serious Adverse Events (SAE) | 321 | 380

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Greater Than or Equal to (>=) Grade 3
Description: Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 (Death) events=death related to an AE.
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 61 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 770 | 784
participants
  Grade 3 or higher TEAE | 405 | 537
  Grade 5 (Death) | 78 | 77

8. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 61 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 770 | 784
participants
  Hypertension | 76 | 98
  Pyrexia | 26 | 41
  Hypotension | 12 | 26

9. Secondary Outcome: Number of Participants With TEAEs Related to Weight
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 61 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 770 | 784
participants
  Weight decreased | 47 | 119
  Weight increased | 36 | 10

10. Secondary Outcome: Number of Participants With Worst Change From Baseline in Eastern Co-operative Oncology Group (ECOG) Performance Status
Description: ECOG assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50 percent of waking hours [hrs]), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50 percent of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Worst change was defined as the worst overall change that occurred in ECOG status at any measured time point during the treatment period.
Time Frame: Baseline until EOT (approximately up to 4.7 years)
Population: Safety population where baseline and post-baseline assessments were available. Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 760 | 771
participants
  Baseline: 0; Overall: 0 | 251 | 200
  Baseline: 0; Overall: 1 | 177 | 237
  Baseline: 0; Overall: 2 | 47 | 66
  Baseline: 0; Overall: 3 | 22 | 15
  Baseline: 0; Overall: 4 | 7 | 7
  Baseline: 1; Overall: 0 | 6 | 6
  Baseline: 1; Overall: 1 | 162 | 147
  Baseline: 1; Overall: 2 | 57 | 60
  Baseline: 1; Overall: 3 | 28 | 26
  Baseline: 1; Overall: 4 | 2 | 6
  Baseline: 2; Overall: 2 | 1 | 1

11. Secondary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings
Time Frame: Baseline up to EOT (Cycle 61 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 770 | 784
participants | 130 | 163

12. Secondary Outcome: Worst Change From Baseline Over Time in Cardiac Ejection Fraction
Description: Worst change was defined as the worst overall change that occurred in cardiac ejection fraction at any measured time point.
Time Frame: Baseline up to 30 days or EOT whichever is later (approximately up to Cycle 61 Day 58)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 676 | 670
percent ejection fraction | -3.8 (6.93) | -4.8 (7.00)

13. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations Related to Chemistry, Hematology or Coagulation
Time Frame: Baseline up to 30 days or EOT whichever is later (approximately up to Cycle 61 Day 58)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 770 | 784
participants
  Investigations | 215 | 399
  Blood and lymphatic system disorders | 114 | 107
  Metabolism and nutrition disorders | 204 | 336

14. Secondary Outcome: Percentage of Participants With Skeletal Related Events (SRE)
Description: Skeletal related (SRE) event is defined as a fracture or spinal cord compression or the need for radiation or surgery at the site of a prostate cancer metastatic lesion that is substantiated by radiographic or pathologic evidence.
Time Frame: Baseline up to EOT (approximately up to 4.7 years)
Population: The ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
percentage of participants | 10.9 [8.8 to 13.3] | 8.6 [6.7 to 10.8]

15. Secondary Outcome: Time to SRE
Description: Time to SRE is defined as the time from randomization to SRE, or death due to any cause, whichever comes first. SRE is defined as a fracture or spinal cord compression or the need for radiation or surgery at the site of a prostate cancer metastatic lesion that is substantiated by radiographic or pathologic evidence.
Time Frame: Baseline up to EOT (Cycle 61 Day 58)
Population: The ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 9.0 [8.32 to 10.98] | 13.9 [13.68 to 16.57]

16. Secondary Outcome: Percentage of Participants Achieving PSA50 Response at Any Time During the Study
Description: The PSA50 is defined as a decline of PSA by 50 percent from baseline.
Time Frame: Cycle: 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34 and 37
Population: ITT population where baseline and post-baseline assessments were available. The ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
percentage of participants
  Cycle 4 (n= 687, 672) | 28.09 [24.76 to 31.62] | 49.70 [45.86 to 53.55]
  Cycle 7 (n= 541, 540) | 34.94 [30.92 to 39.12] | 54.81 [50.51 to 59.07]
  Cycle 10 (n= 438, 450) | 36.99 [32.45 to 41.70] | 56.00 [51.28 to 60.64]
  Cycle 13 (n= 344, 382) | 37.21 [32.09 to 42.56] | 53.14 [48.00 to 58.24]
  Cycle 16 (n= 286, 303) | 34.27 [28.78 to 40.08] | 54.13 [48.33 to 59.84]
  Cycle 19 (n= 228, 272) | 37.72 [31.41 to 44.36] | 52.94 [46.82 to 59.00]
  Cycle 22 (n= 184, 211) | 33.15 [26.40 to 40.46] | 54.03 [47.05 to 60.89]
  Cycle 25 (n= 109, 119) | 35.78 [26.83 to 45.53] | 46.22 [37.04 to 55.59]
  Cycle 28 (n= 67, 77) | 44.78 [32.60 to 57.42] | 48.05 [36.52 to 59.74]
  Cycle 31 (n= 35, 39) | 34.29 [19.13 to 52.21] | 48.72 [32.42 to 65.22]
  Cycle 34 (n= 22, 18) | 36.36 [17.20 to 59.34] | 38.89 [17.30 to 64.25]
  Cycle 37 (n= 7, 5) | 71.43 [29.04 to 96.33] | 40.00 [5.27 to 85.34]

17. Secondary Outcome: Percentage of Participants Achieving 90 Percent Reduction From Baseline in Prostate Specific Antigen (PSA90 Response) at Week 12
Description: The PSA90 is defined as a decline of PSA by 90 percent from baseline.
Time Frame: Week 12
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
percentage of participants | 5.4 | 16.7

18. Secondary Outcome: Percentage of Participants Achieving PSA90 Response at Any Time During the Study
Description: The PSA90 is defined as a decline of PSA by 90 percent from baseline.
Time Frame: Cycle: 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34 and 37
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
percentage of participants
  Cycle 4 (n= 687, 672) | 5.39 [3.82 to 7.35] | 16.67 [13.93 to 19.70]
  Cycle 7 (n= 541, 540) | 8.69 [6.45 to 11.39] | 22.22 [18.78 to 25.97]
  Cycle 10 (n= 438, 450) | 11.64 [8.79 to 15.02] | 26.44 [22.42 to 30.78]
  Cycle 13 (n= 344, 382) | 12.79 [9.45 to 16.79] | 26.18 [21.84 to 30.89]
  Cycle 16 (n= 286, 303) | 12.24 [8.67 to 16.61] | 25.74 [20.91 to 31.05]
  Cycle 19 (n= 228, 272) | 12.72 [8.69 to 17.75] | 26.10 [20.99 to 31.75]
  Cycle 22 (n= 184, 211) | 10.87 [6.77 to 16.29] | 28.44 [22.45 to 35.03]
  Cycle 25 (n= 109, 119) | 11.01 [5.82 to 18.44] | 21.01 [14.08 to 29.43]
  Cycle 28 (n= 67, 77) | 16.42 [8.49 to 27.48] | 27.27 [17.74 to 38.62]
  Cycle 31 (n= 35, 39) | 8.57 [1.80 to 23.06] | 12.82 [4.30 to 27.43]
  Cycle 34 (n= 22, 18) | 4.55 [0.12 to 22.84] | 22.22 [6.41 to 47.64]
  Cycle 37 (n= 7, 5) | 14.29 [0.36 to 57.87] | 20.00 [0.51 to 71.64]

19. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as time from randomization to a PSA increase of 25 percent and PSA rise of at least 2 nanogram per milliliter (ng/mL) above the lowest value observed post baseline or, if no PSA decline occurred post baseline, compared to baseline PSA.
Time Frame: Baseline until the final on treatment assessment or until end of short term follow-up following discontinuation of treatment, whichever occurred later (approximately up to 4.7 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 5.59 [5.56 to 5.59] | 8.3 [8.28 to 8.35]

20. Secondary Outcome: Time to Docetaxel Chemotherapy
Description: Time to docetaxel based chemotherapy is defined as the time from randomization to the start of docetaxel based chemotherapy for prostate cancer, regardless of whether the participant received concurrent orteronel or not. Deaths due to disease progression prior to Docetaxel based chemotherapy were considered as events.
Time Frame: Baseline until start of docetaxel chemotherapy (up to 4.7 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 19.0 [16.44 to 21.43] | 23.0 [20.71 to 24.65]

21. Secondary Outcome: Time to Subsequent Antineoplastic Therapy
Description: Time to subsequent antineoplastic therapy is defined as the time from randomization to the start of any alternate antineoplastic therapy for prostate cancer. Deaths due to disease progression prior to antineoplastic therapy for prostate cancer are considered as events. Otherwise, time to next therapy is censored at the date of death or the last date the participant was known to be alive or the data cutoff date, whichever is earlier.
Time Frame: Baseline until start of subsequent antineoplastic therapy (up to 4.7 years)
Population: The ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 13.9 [12.16 to 14.86] | 17.2 [15.09 to 18.97]

22. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1. A CR was defined as the disappearance of all target lesions determined by computerized tomography (CT) or MRI. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 millimetre (mm). A PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of longest diameters of non-lymph node lesions and of the short diameter or short axis of lymph nodes.
Time Frame: Baseline until disease progression or death, whichever occurred first (approximately up to 4.7 years)
Population: The Response Evaluation Criteria in Solid Tumors (RECIST) evaluable population included all participants who had measurable disease by RECIST 1.1 at the baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 243 | 236
percentage of participants | 15.2 [11.0 to 20.4] | 34.7 [28.7 to 41.2]

23. Secondary Outcome: Time to Deterioration in Global Health Status
Description: Global health status deterioration is defined as a drop greater than 16 points from the baseline assessment, confirmed at least 3 weeks later, on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core Module 30 (EORTC QLQ-C30) index after the score has been linearly transformed to a 0 to 100 scale. EORTC QLQ-C30 consists of 30 questions, where question 1 to 28 can be answered with 1: Not at all, 2: A little, 3: Quite a bit, 4: Very much and question 29 to 30 with 1: Very poor to 7: Excellent. For subscales a high score from 0-100 indicates: high global quality of life, high level of functioning (physical, role, emotional, cognitive, social) or a high level of symptoms (fatigue, nausea, pain, dyspnea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties).
Time Frame: Baseline until EOT (approximately up to 4.7 years)
Population: The ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Number analyzed (Participants) | 779 | 781
months | 10.7 [8.97 to 11.11] | 8.3 [7.36 to 10.16]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to Cycle 61 Day 58).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo + Prednisone 5 mg | Orteronel 400 mg + Prednisone 5 mg
Serious Adverse Events (participants affected / at risk) | 321/770 | 380/784
Other Adverse Events (participants affected / at risk) | 721/770 | 757/784
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Prednisone 5 mg (N=770) | Orteronel 400 mg + Prednisone 5 mg (N=784)
Pneumonia (Infections and infestations) | 9 | 30
Lobar pneumonia (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Bronchopneumonia (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 12
Urosepsis (Infections and infestations) | 4 | 6
Septic shock (Infections and infestations) | 2 | 3
Bacteraemia (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 13
Pyelonephritis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 4 | 3
Appendicitis perforated (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 4
Arthritis bacterial (Infections and infestations) | 0 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 4
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4
Gastroenteritis viral (Infections and infestations) | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 3
Intervertebral discitis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Borrelia infection (Infections and infestations) | 1 | 0
Tongue abscess (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 3 | 9
Diarrhoea (Gastrointestinal disorders) | 5 | 12
Abdominal pain (Gastrointestinal disorders) | 2 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 5
Pancreatitis (Gastrointestinal disorders) | 0 | 4
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 7
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 3
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Gallstone ileus (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 3 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 24
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 12
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to biliary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to urinary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 7
Myocardial infarction (Cardiac disorders) | 5 | 5
Angina pectoris (Cardiac disorders) | 4 | 4
Angina unstable (Cardiac disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 2 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 18 | 14
Atrial flutter (Cardiac disorders) | 3 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 3
Atrial tachycardia (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 7 | 8
Cardiac failure acute (Cardiac disorders) | 3 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 2 | 2
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Cardiomegaly (Cardiac disorders) | 0 | 1
Ventricular hypertrophy (Cardiac disorders) | 0 | 1
Cardiotoxicity (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 23 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal pouch (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 9
Renal failure (Renal and urinary disorders) | 3 | 7
Renal impairment (Renal and urinary disorders) | 0 | 3
Postrenal failure (Renal and urinary disorders) | 2 | 2
Renal injury (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 20 | 13
Urinary hesitation (Renal and urinary disorders) | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 16 | 8
Hydronephrosis (Renal and urinary disorders) | 6 | 5
Obstructive uropathy (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 3 | 3
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Hydroureter (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Urinary bladder rupture (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 5
Cerebral ischaemia (Nervous system disorders) | 2 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 7
Somnolence (Nervous system disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 11 | 6
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 0 | 1
Nerve root compression (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 0 | 2
Paraplegia (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Polyneuropathy (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 2 | 0
IIIrd nerve disorder (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 2 | 11
Asthenia (General disorders) | 1 | 3
Malaise (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 6 | 9
Multi-organ failure (General disorders) | 3 | 3
Multi-organ disorder (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 6
Non-cardiac chest pain (General disorders) | 1 | 4
Discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 2
Face oedema (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Abasia (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 11
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 8
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 5
Pathological fracture (Musculoskeletal and connective tissue disorders) | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 9
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 4
Hypovolaemic shock (Vascular disorders) | 0 | 2
Shock (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 2
Femoral artery occlusion (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 2 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Lipase increased (Investigations) | 5 | 7
Amylase increased (Investigations) | 2 | 2
Pancreatic enzymes increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 2
Liver function test abnormal (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 6
Ejection fraction decreased (Investigations) | 1 | 2
International normalised ratio increased (Investigations) | 1 | 2
Blood calcium increased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 3
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 2
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 | 0
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 18 | 18
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 4
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 2
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1
Thyrotoxic crisis (Endocrine disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Allergy to arthropod sting (Ear and labyrinth disorders) | 0 | 1
Drug hypersensitivity (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Prednisone 5 mg (N=770) | Orteronel 400 mg + Prednisone 5 mg (N=784)
Anaemia (Blood and lymphatic system disorders) | 90 | 75
Nausea (Gastrointestinal disorders) | 130 | 281
Constipation (Gastrointestinal disorders) | 129 | 261
Diarrhoea (Gastrointestinal disorders) | 110 | 221
Vomiting (Gastrointestinal disorders) | 115 | 174
Abdominal pain (Gastrointestinal disorders) | 40 | 72
Dyspepsia (Gastrointestinal disorders) | 33 | 60
Abdominal pain upper (Gastrointestinal disorders) | 39 | 51
Fatigue (General disorders) | 173 | 269
Asthenia (General disorders) | 70 | 106
Oedema peripheral (General disorders) | 85 | 86
Urinary tract infection (Infections and infestations) | 60 | 58
Fall (Injury, poisoning and procedural complications) | 47 | 57
Lipase increased (Investigations) | 35 | 179
Weight decreased (Investigations) | 54 | 124
Amylase increased (Investigations) | 27 | 146
Blood creatinine increased (Investigations) | 21 | 78
Alanine aminotransferase increased (Investigations) | 14 | 49
Decreased appetite (Metabolism and nutrition disorders) | 86 | 170
Diabetes mellitus (Metabolism and nutrition disorders) | 23 | 45
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 47
Dehydration (Metabolism and nutrition disorders) | 18 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 196 | 158
Muscle spasms (Musculoskeletal and connective tissue disorders) | 118 | 171
Arthralgia (Musculoskeletal and connective tissue disorders) | 122 | 123
Pain in extremity (Musculoskeletal and connective tissue disorders) | 93 | 79
Bone pain (Musculoskeletal and connective tissue disorders) | 75 | 65
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 64 | 55
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 42 | 51
Muscular weakness (Musculoskeletal and connective tissue disorders) | 42 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 45
Dizziness (Nervous system disorders) | 50 | 105
Headache (Nervous system disorders) | 50 | 70
Dysgeusia (Nervous system disorders) | 15 | 46
Insomnia (Psychiatric disorders) | 65 | 84
Depression (Psychiatric disorders) | 23 | 56
Haematuria (Renal and urinary disorders) | 45 | 43
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 | 84
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 62
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 22 | 41
Hypertension (Vascular disorders) | 80 | 98
Hot flush (Vascular disorders) | 77 | 81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.